CLINICAL TRIAL: NCT00345852
Title: A Prospective, Randomized Multicenter Trial of Amnioreduction Vs Selective Fetoscopic Laser Photocoagulation for the Treatment of Severe Twin-Twin Transfusion Syndrome
Brief Title: Fetoscopic Selective Laser Photocoagulation in Twin-Twin Transfusion Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HD041149 (NIH); NCT00109694 (obsolete NCT alias)
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2007-06-29 (Estimated); Status verified 2006-06

CONDITIONS: Twin to Twin Transfusion Syndrome
Keywords: twin to twin transfusion syndrome; fetoscopic selective laser photocoagulation; amnioreduction
MeSH Terms: conditions — Fetofetal Transfusion

INTERVENTIONS:
Procedure: Fetoscopic Selective Laser Photocoagulation

SUMMARY:
This is a study to compare two treatments (amnioreduction vs. selective fetoscopic laser photocoagulation [SFLP]) in patients with severe twin to twin transfusion syndrome.

DETAILED DESCRIPTION:
We hypothesize that treatment of the underlying chorioangiopagus by selective fetoscopic laser photocoagulation will not only improve the survival of twins but will reduce the incidence of neurologic, cardiac, and developmental sequelae of twin-twin transfusion syndrome (TTTS). We propose to test this hypothesis by a prospective randomized multicenter trial to compare serial amnioreduction with selective fetoscopic laser photocoagulation in cases of severe (stage II-IV) twin-twin transfusion syndrome (TTTS). Primary Outcomes: Survival of donor twin at 30 days after birth and no treatment failure; Survival of recipient twin at 30 days after birth and no treatment failure; Secondary Outcomes: Survival times of each twin in utero or after birth (which may be censored at 30 days after birth); Gestational age at delivery; Placental insufficiency; Cardiac outcome: echocardiographic evidence of cardiac compromise; Neurologic outcome: evidence of brain injury preceding birth by MRI; Postnatal comorbidity

ELIGIBILITY:
Inclusion Criteria:

* Both twins are alive
* TTTS diagnosed prior to 22 weeks gestation
* Monochorionic diamniotic gestation
* Like sex twins
* Single placental mass
* Thin intertwin membrane
* Oligohydramnios in donor twin (deepest vertical pocket of ≤ 2 cm)
* Polyhydramnios with deepest vertical pocket of > 8 cm with or without Doppler or echocardiographic changes in the recipient twin (deepest vertical pocket of > 6 cm if previous amnioreduction)
* Decompressed bladder in donor not seen to fill during the ultrasound examination (stage II, III, or IV), unless Doppler velocimetry changes (absent end-diastolic umbilical artery flow, abnormal ductus venosus waveform), and/or echocardiographic changes (valvular insufficiency, ventricular hypertrophy) are already present
* No associated structural abnormalities
* No sonographic evidence of CNS injury at time of entry
* No preterm labor
* No maternal medical contraindication to anesthesia or surgery

Exclusion Criteria:

* Failure to meet all inclusion criteria
* TTTS presenting after 22 weeks gestation
* Randomization after 24 weeks gestation
* Cervical length < 2.0 cm post initial
* Presence of cervical cerclage
* Uterine anomaly
* Refusal to accept randomization
* Unable to pursue prenatal care at an approved center coordinated by one of the participating institutions
* Unable to pursue postnatal evaluation at a NICHD Neonatal Research Network Institution

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-03; Study Completion 2007-05

PRIMARY OUTCOMES:
Survival of donor twin at 30 days after birth and no treatment failure
Survival of recipient twin at 30 days after birth and no treatment failure

SECONDARY OUTCOMES:
Survival times of each twin in utero or after birth (which may be censored at 30 days after birth)
Gestational age at delivery
Placental insufficiency
Cardiac outcome: echocardiographic evidence of cardiac compromise
Neurologic outcome: evidence of brain injury preceding birth by MRI
Postnatal comorbidity

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Crombleholme, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (12):
- United States (12):
  - University of California-San Francisco, San Francisco, California
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - New York University School of Medicine, New York, New York
  - Columbia-Presbyterian Medical Center, New York, New York
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Magee-Women's Hospital, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- See also: Fetal Care Center of Cincinnati Twin-Twin Transfusion Syndrome (TTTS) webpage — http://www.fetalcarecenter.org/medicine/therapies/ttts/